CLINICAL TRIAL: NCT07102563
Title: Investigating the Biological Link Between Mental Health Status and Outcomes Following Total Knee and Hip Replacement.
Brief Title: Biological Link Between Anxiety and Outcomes Post Knee Arthroplasty
Status: Not yet recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 914
Record Dates: First submitted 2025-07-30; First posted 2025-08-03 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TKR patients with anxiety/depression (14): TKR patients with anxiety/depression (14)
- TKR patients without anxiety/depression (14): TKR patients without anxiety/depression (14)
- THR patients with anxiety/depression (14): THR patients with anxiety/depression (14)
- THR patients without anxiety/depression (14): THR patients without anxiety/depression (14)

SUMMARY:
This is a single-site, observational pilot study that aims to understand whether there is a biological explanation for why some patients with anxiety or depression experience poorer outcomes after total knee or hip replacement surgery. The study investigates the role of inflammation inside the joint, using tissue, fluid, and blood samples collected during routine care, alongside patient-reported outcome questionnaires.

Study Design and Hypothesis The hypothesis is that patients with pre-existing anxiety or depression will show more inflammation in their joint tissue or blood, and that this may be linked to poorer functional outcomes after surgery. An alternative explanation is that these patients may report worse outcomes without an identifiable biological cause.

The study does not involve any trial drugs or new treatments and does not use a placebo or randomisation.

Patients will be grouped based on whether or not they meet the criteria for anxiety and/or depression as measured by two validated mental health screening tools:

GAD-7 (for anxiety)

PHQ-8 (for depression)

Sampling and Participant Involvement:

The plan is to include 56 patients, equally split between hip and knee replacement groups, and between those with and without anxiety/depression (14 per subgroup). Participants will be identified by the clinical research team from the waiting lists of two lead surgeons and approached by post and phone before their routine preoperative assessment clinic.

At that appointment, consent will be obtained and the participant will complete baseline questionnaires. The same questionnaires will be repeated at 3 and 6 months postoperatively. No additional visits will be required.

Study Procedures and Timeline

1. Preoperative phase (routine clinic visit):

   Participants are posted a cover letter, patient information sheet, and consent form ahead of their clinic visit.

   A member of the research team calls the patient to explain the study.

   At the clinic, a research nurse obtains informed consent.

   Participants complete baseline questionnaires assessing pain, quality of life, and mental wellbeing (e.g. Oxford score, EQ-5D, PHQ-8, GAD-7).
2. Day of surgery:

   An additional 20 ml of blood is collected at the same time as routine preoperative blood tests, using the same venepuncture.

   While under anaesthetic, the operating surgeon collects small tissue samples (synovial fluid, synovial tissue, and fat) from the joint. These samples are normally discarded as part of the operation.

   Samples are anonymised and sent to pathology and research laboratories for analysis.
3. Postoperative follow-up:

At the 3-month clinic visit (routine care), participants complete the same questionnaires and provide a further blood sample of approximately 15 ml.

At 6 months, questionnaires are completed remotely via the MyRecovery app, with no further hospital visit or samples required.

All study procedures are aligned with routine NHS care to minimise burden. There are no additional clinic visits required.

Data Handling and Analysis The study will compare inflammation levels (in blood and tissue) between groups and analyse how these relate to patient-reported outcomes. All data will be anonymised. Blood samples will be processed at local NHS labs (Shrewsbury) and at a specialist centre in Sheffield for specific inflammatory markers (e.g. IL-6, CD solubles). Synovial tissue will be histologically analysed on-site for synovitis.

DETAILED DESCRIPTION:
This study aims to investigate the potential biological mechanisms linking preoperative anxiety and depression with poorer patient-reported outcomes following total knee or hip replacement surgery. Specifically, we are exploring whether psychological distress is associated with increased local joint inflammation (synovitis) and whether this may mediate reduced functional recovery. Biological samples (including synovial fluid, synovial tissue, and fat pad) will be collected intraoperatively from routine surgical waste, and additional blood samples will be analysed for routine blood tests (FBC, Renal function tests, Liver function tests) and inflammatory markers (CRP, ESR, IL-6, CD solubles). We will correlate these findings with validated psychological and functional outcome measures collected pre- and postoperatively.

Recruitment and Consent:

Patients scheduled for elective knee or hip replacement at the Robert Jones and Agnes Hunt Orthopaedic Hospital will be screened for eligibility by a clinician as part of the care team. Eligible patients will receive a patient information sheet and consent form by post ahead of their routine preoperative clinic visit. A telephone call will follow to confirm interest. Final written informed consent will be obtained by a trained research nurse at the preoperative assessment clinic. Participants may decline or withdraw from the study at any time without affecting their standard clinical care.

Risks, Burdens, and Benefits:

The risks associated with participation are minimal. All tissue samples will be collected during routine surgery while the patient is under general anaesthesia, using tissue that would otherwise be discarded. A small additional blood sample (20 ml) will be collected on the day of surgery using the same venepuncture as for routine bloods, and a follow-up sample (approx. 15 ml) will be withdrawn at the routine 3-month clinic visit. The risks of blood withdrawal are minimal such as discomfort or bruising. However, a senior trained staff will withdraw all the blood tests to minimise any potential risks. Questionnaires on anxiety and depression might cause mild emotional discomfort; appropriate safeguarding procedures are in place, and GP referrals will be made for participants scoring above clinical thresholds. Participants will be informed of their blood test results related to inflammation, where clinically appropriate.

Confidentiality and Data Security:

All identifiable information will be stored securely, in accordance with the Data Protection Act 1998 and current NHS policies. Each participant will be assigned a unique study ID. Identifiable data will be kept separate from research data and stored in encrypted, password-protected files. Only authorised research staff will have access. Biological samples sent for external analysis (IL-6 and CD solubles in Sheffield Hospital) will be fully anonymised.

Use and Storage of Samples:

The institution holds appropriate approvals under the Human Tissue Act to store and use human biological samples. Any remaining samples may be stored securely in the RJAH Arthritis Research Centre laboratory for future ethically approved research. No genetic testing will be performed. Samples may be transported to partner laboratories within the UK for specific assays, using NHS-compliant logistics.

Ethical and Organisational Oversight:

This is a single-site, low-risk observational study embedded within routine NHS care. There are no additional clinic visits or interventions. Ethical, data protection, and sample handling issues have been reviewed and addressed through standard NHS research governance procedures, and the study has received peer review and 'agreement in principle' from all relevant support departments.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Scheduled to undergo elective total knee replacement (TKR) or total hip replacement (THR) at the Robert Jones and Agnes Hunt Orthopaedic Hospital.
3. Body mass index (BMI) less than 35

Exclusion Criteria:

1. Rheumatoid arthritis or inflammatory arthropathies.
2. Patients on Steroids, Aspirin, or Cox inhibitors.
3. Smokers or vapers.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total knee replacement (TKR) or total hip replacement (THR) patients.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
The correlation between preoperative anxiety and/or depression following total knee replacement (TKR) versus total hip replacement (THR). | For the first 6 months following TKR or THR surgery.
  The primary outcome measure is the correlation between preoperative anxiety and/or depression (measured by validated mental health questionnaires) and postoperative outcomes (measured by patient-reported outcome measures, or PROMs) following total knee replacement (TKR) versus total hip replacement (THR).
  Specifically, the study will assess:
  Whether the severity of anxiety or depression is associated with worse PROMs (e.g. Oxford Knee or Hip Score, EQ-5D) at 3 and 6 months after surgery.
  Whether this relationship is influenced (mediated) by the presence and severity of synovitis (joint inflammation) and inflammatory cytokines (measured in synovial fluid and blood).

SECONDARY OUTCOMES:
Correlation between preoperative anxiety/depression , synovitis grade and inflammatory markers in synovial fluid with systemic inflammation. | For the first 6 months following TKR or THR surgery.
  Blood biomarkers such as CRP, ESR, IL-6, and CD solubles.
  Differences in hospital stay duration, readmission rates, and postoperative complications between:
  Patients who report satisfaction versus dissatisfaction after surgery, and Patients with versus without preoperative anxiety/depression, stratified by joint type (total knee replacement vs total hip replacement).

CONTACTS AND LOCATIONS:
Locations (1):
- The Robert Jones and Agnes Hunt Orthopaedic Hospital, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blackburn J, Qureshi A, Amirfeyz R, Bannister G. Does preoperative anxiety and depression predict satisfaction after total knee replacement? Knee. 2012 Oct;19(5):522-4. doi: 10.1016/j.knee.2011.07.008. Epub 2011 Aug 16. PMID 21846588
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Nam D, Nunley RM, Barrack RL. Patient dissatisfaction following total knee replacement: a growing concern? Bone Joint J. 2014 Nov;96-B(11 Supple A):96-100. doi: 10.1302/0301-620X.96B11.34152. PMID 25381418
- [Background] Scott CE, Howie CR, MacDonald D, Biant LC. Predicting dissatisfaction following total knee replacement: a prospective study of 1217 patients. J Bone Joint Surg Br. 2010 Sep;92(9):1253-8. doi: 10.1302/0301-620X.92B9.24394. PMID 20798443
- [Background] DeFrance MJ, Scuderi GR. Are 20% of Patients Actually Dissatisfied Following Total Knee Arthroplasty? A Systematic Review of the Literature. J Arthroplasty. 2023 Mar;38(3):594-599. doi: 10.1016/j.arth.2022.10.011. Epub 2022 Oct 14. PMID 36252743
- [Background] Anakwe RE, Jenkins PJ, Moran M. Predicting dissatisfaction after total hip arthroplasty: a study of 850 patients. J Arthroplasty. 2011 Feb;26(2):209-13. doi: 10.1016/j.arth.2010.03.013. Epub 2010 May 11. PMID 20462736
- [Background] Versus Arthritis. Tackling osteoarthritis - the UK's leading cause of pain and disability. Versus Arthritis. 2021.